CLINICAL TRIAL: NCT03416361
Title: VItamiN D treatIng Chronic heArT Failure (the Effect of Vitamin D Supplementation on Hospitalisation and Mortality in Patients With Heart Failure): Multicentre, Phase III, Randomised Placebo-controlled Trial
Brief Title: VItamiN D treatIng Chronic heArT Failure (the Effect of Vitamin D Supplementation in Patients With Heart Failure)
Acronym: VINDICATE2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, KK Witte, Senior Lecturer in Cardiology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 224168
Record Dates: First submitted 2017-12-04; First posted 2018-01-31 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Chronic Heart Failure
Keywords: Left ventricular dysfunction; Vitamin D
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): 4000IU Vitamin D3 as two 50mcg tablets per day
  Interventions: Dietary Supplement: 4000IU Vitamin D3
- Control (Placebo Comparator): Placebo - two chewable blackcurrant flavoured tablets per day
  Interventions: Dietary Supplement: 4000IU Vitamin D3

INTERVENTIONS:
Dietary Supplement: 4000IU Vitamin D3 — Chewable blackcurrant flavoured tablets (two per day)

SUMMARY:
VINDICATE 2 will be a randomised, placebo-controlled, parallel group, double-blind study of vitamin D versus placebo in otherwise optimally-managed patients with CHF due to LVSD and vitamin D deficiency (<50nmol/L). The intervention will be a daily dose of 4000IU (100µg) per day or matching placebo for a minimum of 2 years and a maximum of 4 years.

DETAILED DESCRIPTION:
DESIGN: Multi-centre, phase III, double-blind, parallel-group, placebo-controlled trial.

SETTING: Secondary care heart failure clinics across the UK. TARGET POPULATION: Higher-risk patients with CHF due to LVSD recruited from CHF clinics.

HEALTH TECHNOLOGY: 4000IU (100mcg) vitamin D3 or placebo daily for minimum 2yrs and maximum 4yrs.

MEASUREMENT OF OUTCOMES:

Primary end-point is a composite of HF hospitalisation or death Secondary outcomes include all-cause mortality, hospitalisations and cost-effectiveness. Patient outcomes will be obtained from NHS Digital (KKW is an approved researcher) with a transfer of linked data to be held at the Leeds Institute for Data Analysis.

Patient reported outcomes will be Minnesota Living with HF questionnaire and EQ-5D which will be assessed at twelve-monthly research visits.

SAMPLE SIZE: Based on VINDICATE, 2-yr CV mortality or hospitalisation in stable high-risk HF is 28% in those receiving placebo and 21% in those receiving vitamin D3 (hazard ratio 0.717). In the largest observational study (n=1800) of the effect of vitamin D deficiency on outcomes in patients with CHF on optimal medical therapy, balanced for all important variables except vitamin D, there was a significant adverse effect of vitamin D deficiency on all-cause mortality, demonstrating a 14% reduction in death for each 2.72-fold increase in vitamin D.

To demonstrate this effect 379 events in 1278 patients are required. Calculations assume time to CV event follows an exponential distribution, 2-sided 5% level of significance, 90% power, 20% dropout, 2.5-yrs recruitment and min. 2-yr follow-up.

ANALYSIS: Primary analysis will be on an intention-to-treat basis. Cox proportional hazards regression will be fitted to the time to first CV event adjusted for stratification factors.

Health Economics: A model will estimate lifetime incremental costs from an NHS/PSS perspective and QALYs gained based data from VINDICATE-2 and the literature. ICERs will be estimated and compared to standard cost-effectiveness thresholds to determine if vitamin D3 supplementation is cost-effective. Further analyses will explore the value of investing in activities to support uptake of vitamin D3 in clinical practice.

CURRENT AND PLANNED CARE PATHWAYS: The pathway within the study will be 4000IU vitamin D3 daily or placebo followed by safety and adherence visits at 3m and 12 monthly post-randomisation up to final visit at 24-48m. Patients will be screened, recruited and followed up during standard clinic visits. A small parcel containing three months of the intervention will be posted to participants by Leeds Teaching Hospitals Pharmacy every three months for the duration of their involvement in the study.

If adopted into standard care pathways, vitamin D could be prescribed and monitored cheaply and easily in primary care with annual blood tests.

PROJECT TIMETABLES: Set-up 6m, recruitment 30m, follow-up 24m, data cleaning, analysis and reporting 6m - total 66m.

RECRUITMENT RATE: 5 main centres (+2 PIC sites), 3.55 pts/mth/centre.

ELIGIBILITY:
Inclusion Criteria:

* LVSD (LVEF <50%);
* stable medical and device therapy for >3mths;
* 25[OH]vitamin D3 <50nmol/L
* At least one of: recent (<1 year) hospitalisation for HF, high dose loop diuretic requirement (>80mg daily furosemide equiv), diabetes mellitus, ischaemic aetiology

Exclusion Criteria:

* Unwilling/unable to sign consent,
* Severe cognitive impairment,
* Severe COPD,
* Anaemia,
* Other life-threatening co-morbidity (in the opinion of the local co-investigator),
* Known and active sarcoidosis or tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1253 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Combined heart failure hospitalisation and total mortality | 24 months
  Time to death or first hospitalisation for heart failure

SECONDARY OUTCOMES:
Total mortality | 24 months
  Time to death
Cost effectiveness | 24 months
  ICER for vitamin D
Change in patient quality of life | 24 months
  EQ5D - 5L

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data to be made available from the Leeds Institute of Data Analytics